CLINICAL TRIAL: NCT04130828
Title: Thrice-weekly Versus Thrice-daily Oral Ferrous Fumarate Treatment in Adult Patients With Iron Deficiency Anemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Collaborators: The Thai Society of Hematology (Unknown)
Responsible Party: Principal Investigator, Siddhibhong Jongkraijakra, Faculty of Pharmaceutical scienes, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC.62-404-14-1
Record Dates: First submitted 2019-10-16; First posted 2019-10-17 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Iron Deficiency Anemia
Keywords: ferrous fumarate; oral iron treatment; thrice-weekly; thrice-daily; iron deficiency anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thrice-weekly group (Experimental): Ferrous fumarate 200 mg PO PC Thrice-weekly
  Interventions: Drug: Ferrous Fumarate
- Thrice-daily group (Active Comparator): Ferrous fumarate 200 mg PO PC Thrice-daily
  Interventions: Drug: Ferrous Fumarate

INTERVENTIONS:
Drug: Ferrous Fumarate — Ferrous fumarate 200 mg PO PC

SUMMARY:
Iron deficiency anemia is a global health problem and the most common cause of anemia worldwide. Patients with iron deficiency and Iron deficiency anemia can present with a multitude of symptoms including fatigue, dyspnea on exertion, dysphagia, pallor, palpitations, headaches, tinnitus, taste disturbance and pica. Oral iron supplementation is associated with increasing hemoglobin in multiple studies in women, pregnant women and elderly patients. However, the optimal dose and frequency of oral iron supplementation for treatment remains unclear. The current proposed study attempts to address this gap in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients with iron deficiency anemia defined as hemoglobin less than 12 g/dL in women or 13 g/dL in men; AND ferritin less than 30 ng/mL

Exclusion Criteria:

* Allergy to iron
* Currently pregnancy
* Currently breastfeeding
* Known history of inflammatory bowel disease, celiac disease, inherited bleeding disorder, solid cancer, hematologic cancer or thalassemia
* Renal impairment or glomerular filtration rate less than 30 ml/min/1.73m2
* Hepatic impairment or Child Pugh score more than 7
* Active bleeding define hemoglobin decrease more than 2 g/dL
* Multivitamin and mineral supplement (35 mg or more of elemental iron per day) in 2 weeks prior to randomization
* Non-literate

Subject withdrawal criteria:

* Intolerance to drugs
* Active bleeding define hemoglobin decrease more than 2 g/dL
* Major surgery
* Blood transfusion
* Loss follow-up more than 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-01-21 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Proportion of patient who achieved hemoglobin target | 12 weeks
  Hemoglobin achieved 12 g/dL in women, 13 g/dL in men and or increased 1g/dL/4weeks

SECONDARY OUTCOMES:
Safety and Tolerability: Incidence of Treatment-Emergent Adverse Events | 12 weeks
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Songklanagarind Hospital, Hat Yai, Changwat Songkhla, Thailand

IPD SHARING:
Plan to Share IPD: No